CLINICAL TRIAL: NCT01755039
Title: Verlauf Und Respiratorische Zwischenfälle Bei Patienten Mit außerklinischer Beatmung
Brief Title: Course and Complications of Invasive Out-of-hospital Ventilation
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Other Study IDs: WI_Heimbeatmung_61/2009
Record Dates: First submitted 2012-03-09; First posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Indication for Invasive Out-of-hospital Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with invasive out-of-hospital ventilation

SUMMARY:
The purpose of the study is to determine the frequency and management of respiratory incidence in patients with invasive out-of-hospital ventilation, either living at home for elderly people allay to a weaning centre or at home. Further, the mortality and the frequency of hospital admission will be analyzed.

DETAILED DESCRIPTION:
Background: There has been arise in a number of patients requiring long term ventilation both in the in-hospital as well as the out-of-hospital setting. Despite this, little is known about the subsequent political course of this patients following hospital discharge.

Interventions: This is an observational prospective study over a period of one year in a sample of 50 to 70 invasively ventilated patients living either in a nursing home specialized in the care of ventilated patients or at home. Protocol had been developed containing 20 suspected emergency incidences in respiratory care. The nursing staffs are instructed about the study and how to complete the protocol. The protocol was placed at each patient and every time an emergency occurred, the nursing staff registered the incidence. If an emergency fulfils more than one criterion in the protocol, every applicable criterion was marked. The data will be analyzed using non-parametric descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* existing out-of-hospital ventilation >6h in 24h

Exclusion Criteria:

* Age <18 years
* absence of declaration of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for out-of-hospital ventilation
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Respiratory Incidences | Over a 12-month period, monthly
  Incidences comprise:
  permanent alarming by the ventilator, malfunction of the ventilator, use of an AMBU bag, dyspnoea, worsening of general condition, desaturation of 5 % or more in relation to average saturation of the patients, disconnection of the ventilator, increase of tracheal secretion, reanimation, replacement of tracheal canula, other emergency, call of emergency doctor, call of pneumologist, unscheduled home visit of the patient by a doctor, use of antibiotics, use ov steroids, use of opiates, changing of the ventilator settings, hospital transfer, death.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- Wissenschaftliches Institut Bethanien e.V., Solingen, Germany